CLINICAL TRIAL: NCT00484419
Title: Effects of Colesevelam HCl, Avandia® (Rosiglitazone Maleate), or JanuviaTM (Sitagliptin) on Glycemic Parameters and Lipid Profiles in Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin Monotherapy
Brief Title: Effects of Colesevelam HCl, Rosiglitazone, Sitagliptin on Control of Blood Glucose and Lipids in Type 2 Diabetes Patients Whose Blood Glucose Isn't Completely Controlled With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wel-409
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes; Hyperlipidemia
Keywords: Colesevelam HCl,; rosiglitazone; sitagliptin; Type 2 diabetes; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperlipidemias | interventions — Colesevelam Hydrochloride; Rosiglitazone; Sitagliptin Phosphate

ARMS (3):
- colesevelam (Experimental): colesevelam tablets 625 mg
  Interventions: Drug: Colesevelam HCl
- rosiglitazone (Active Comparator): rosiglitazone maleate 4mg
  Interventions: Drug: rosiglitazone maleate
- sitagliptin (Active Comparator): sitagliptin phosphate tablets
  Interventions: Drug: sitagliptin phosphate

INTERVENTIONS:
Drug: Colesevelam HCl — coleveselam tablets 625 mg; 6 tablets/day
  Arms: colesevelam
Drug: rosiglitazone maleate — rosiglitazone tablets 4mg
  Arms: rosiglitazone
Drug: sitagliptin phosphate — sitagliptin phosphate tablets 100mg/day
  Arms: sitagliptin

SUMMARY:
A 16 week open-label study with subjects receiving background metformin monotherapy. 150 subjects randomized 1:1:1 to receive 1 of the following: open-label colesevelam HCl, open label rosiglitazone, or open-label sitagliptin.

ELIGIBILITY:
Inclusion Criteria:

* HbA1C 7.0 % to 10.0% on metformin monotherapy; may be withdrawn from other (non-metformin) drugs if HbA1C is 6.5% to 9.5 % at screening.

Exclusion Criteria:

* Subjects currently treated with a thiazolidinedione are excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - La Mesa, California
  - Los Angeles, California
  - Los Gatos, California
  - San Antonio, California
  - Chiefland, Florida
  - Gary, Indiana
  - Baltimore, Maryland
  - Dearborn, Michigan
  - West Bloomfield, Michigan
  - Las Vegas, Nevada
  - Yonkers, New York
  - Lexington, North Carolina
  - Winston-Salem, North Carolina
  - Munroe Falls, Ohio
  - Zaneville, Ohio
  - Portland, Oregon
  - Jersey Shore, Pennsylvania
  - Clemson, South Carolina
  - Harriman, Tennessee
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 18 May 2007 to 14 December 2007 at 6 sites in Colombia, 7 sites in Mexico, and 20 sites in the United States of America.
Pre-assignment Details: Subjects on metformin-combination therapy entered a 4-week washout period from non-metformin antidiabetic drug. Population is type 2 diabetes mellitus subjects on stable metformin regimen, who discontinued other antidiabetic drugs, glycemia not controlled, and low-density lipoprotein-C (LDL-C) >=60 mg/dL and triglycerides <500 mg/dL
Groups:
- Sitagliptin: sitagliptin phosphate tablets 100mg
Period: Overall Study
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Started | 57 | 56 | 56
Completed | 45 | 51 | 45
Not Completed | 12 | 5 | 11
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — subject met discontinuation criteria | 2 | 2 | 4
Not completed — required restricted medication | 1 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 1
Not completed — subject unable to receive medication | 1 | 0 | 0
Not completed — subject relocated | 0 | 1 | 0
Not completed — sponsor decision, randomized in error | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin | Total
Number analyzed (Participants) | 57 | 56 | 56 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 46 | 135
  >=65 years | 12 | 12 | 10 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.19) | 54.7 (10.92) | 54.8 (9.76) | 55.4 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 36 | 98
  Male | 28 | 23 | 20 | 71
Region of Enrollment [Number; unit: participants]
  Colombia | 21 | 12 | 19 | 52
  Mexico | 12 | 19 | 12 | 43
  United States | 24 | 25 | 25 | 74
Fasting Insulin [Mean (Full Range); unit: uIU/mL] — baseline fasting insulin
  uIU/mL | 9.406 [1.63 to 47.77] | 9.945 [1.22 to 42.37] | 8.886 [1.32 to 24.02] | 9.396 [1.22 to 47.77]
Fasting Plasma Glucose [Mean (Full Range); unit: mg/dL] — baseline Fasting Plasma Glucose (FPG)
  mg/dL | 174.5 [109 to 270] | 177.7 [101 to 469] | 180.6 [85 to 456] | 177.6 [85 to 469]
HbA1c [Mean (Full Range); unit: percent] — baseline glycosylated hemoglobin
  percent | 8.10 [6.8 to 9.7] | 8.06 [6.7 to 9.7] | 8.17 [6.5 to 9.9] | 8.11 [6.5 to 9.9]

OUTCOME MEASURES:

1. Secondary Outcome: Mean Percentage of Change in Glycosylated Hemoglobin (HbA1c) From Week 0(Baseline) to Week 16 Endpoint Least Squares Mean
Description: Change in HbA1c from Week 0(baseline)to Week 16 endpoint least squares mean with 95% confidence intervals, change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: The Full Analysis Set population included all randomized subjects who had taken at least 1 dose of study medication, and had a baseline and at least 1 post baseline HbA1c measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in HbA1c
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 56 | 54 | 55
% change in HbA1c | -0.27 [-0.52 to -0.02] | -0.58 [-0.83 to -0.32] | -0.38 [-0.64 to -0.13]

2. Secondary Outcome: Mean Percentage of Change in HbA1c From Week 0(Baseline) to Week 8
Description: change in HbA1c from Week 0(baseline) to week 8 mean and standard deviation change = week 8 - week 0.
Time Frame: 8 weeks change = week 8- week 0.
Measure: Mean (Standard Deviation); unit: % change in HbA1c
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 51 | 53 | 48
% change in HbA1c | -0.31 (0.772) | -0.19 (0.842) | -0.48 (0.751)
Statistical Analysis 1: Comparison: Colesevelam; For a treatment group, assuming a within-subject standard deviation of at most 1.15, a 2-sided t-test of the null hypothesis that the change from baseline (CFB) is zero will have 67% to 85% power to detect a difference of 0.4 to 0.5 with a sample size of 50 randomized subjects; Test type: Superiority or Other; p = 0.0061, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1090, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Primary Outcome: Mean Percentage of Change in HbA1c From Week 0(Baseline) to Week 16 Endpoint
Description: Change in HbA1c from Week 0(baseline) to Week 16 endpoint mean with standard deviation change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change HbA1c
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 46 | 51 | 43
% change HbA1c | -0.31 (0.898) | -0.65 (0.836) | -0.56 (1.044)
Statistical Analysis 1: Comparison: Colesevelam; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0234, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0011, t-test, 2 sided

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Week 0(Baseline) to Week 8 Least Squares Mean
Description: change in FPG from Week 0(baseline) to week 8 least squares mean and 95% confidence interval change = week 8 - week 0.
Time Frame: 8 weeks change = week 8- week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 51 | 53 | 48
mg/dL | -15.6 [-25.8 to -5.3] | -28.9 [-38.9 to -18.8] | -17.4 [-28.0 to -6.9]

5. Secondary Outcome: Change in FPG From Week 0(Baseline) to Week 16 Least Squares Mean
Description: change in FPG from Week 0(baseline) to week 16 least squares mean and 95% confidence interval change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 46 | 51 | 45
mg/dL | -17.3 [-28.9 to -5.7] | -31.4 [-42.5 to -20.4] | -24.4 [-36.1 to -12.6]

6. Secondary Outcome: Mean Change in FPG From Week 0(Baseline) to Week 8
Description: mean change in FPG from Week 0(baseline) to Week 8 with standard deviation change = week 8 - week 0.
Time Frame: 8 weeks change = week 8- week 0.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 51 | 53 | 48
mg/dL | -12.5 (32.22) | -30.8 (59.67) | -18.6 (63.56)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0077, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0004, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0483, t-test, 2 sided

7. Secondary Outcome: Mean Change in FPG From Week 0(Baseline) to Week 16
Description: change in FPG from Week 0(baseline) to week 16 mean and standard deviation change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 46 | 51 | 45
mg/dL | -15.8 (41.53) | -34.0 (63.55) | -23.1 (59.49)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0133, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0004, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0125, t-test, 2 sided

8. Secondary Outcome: Change in Fasting Insulin From Week 0(Baseline) to Week 8 Least Squares Mean
Description: change in fasting insulin from Week 0(baseline) to week 8 least squares mean and 95% confidence interval change = week 8 - week 0.
Time Frame: 8 weeks change = week 8- week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: uIU/mL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 48 | 47 | 45
uIU/mL | 0.075 [-3.442 to 3.592] | -2.156 [-5.720 to 1.408] | 4.002 [0.371 to 7.633]

9. Secondary Outcome: Change in Fasting Insulin From Week 0(Baseline) to Week 16 Least Squares Mean
Description: change in fasting insulin from Week 0(baseline) to week 16 least squares mean and 95% confidence interval change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: uIU/mL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 45 | 45 | 44
uIU/mL | -0.320 [-1.757 to 1.116] | -1.482 [-2.922 to -0.041] | 0.092 [-1.363 to 1.547]

10. Secondary Outcome: Mean Change in Fasting Insulin From Week 0(Baseline) to Week 8
Description: mean change in fasting insulin from Week 0(baseline) to week 8 with standard deviation change = week 8 - week 0.
Time Frame: 8 weeks change = week 8- week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 48 | 47 | 45
uIU/mL | 0.107 (4.1543) | -2.213 (6.5833) | 4.028 (20.1202)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.8596, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0257, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.1862, t-test, 2 sided

11. Secondary Outcome: Mean Change in Fasting Insulin From Week 0(Baseline) to Week 16
Description: mean change in fasting insulin from Week 0(baseline) to week 16 with standard deviation change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 45 | 45 | 44
uIU/mL | -0.212 (3.7914) | -1.910 (8.5117) | -0.419 (3.6669)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.7094, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.1394, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.4528, t-test, 2 sided

12. Secondary Outcome: Change in Post-prandial Glucose From Week 0(Baseline) to Week 16 Least Squares Mean
Description: change in post-prandial glucose from Week 0(baseline) to week 16 least squares mean with 95% confidence intervals change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 45 | 48 | 45
mg/dL | -17.7 [-34.8 to -0.7] | -53.6 [-70.1 to -37.1] | -43.6 [-60.7 to -26.6]

13. Secondary Outcome: Mean Change in Post-prandial Glucose From Week 0(Baseline) to Week 16
Description: mean change in post-prandial glucose from Week 0(baseline) to week 16 with standard deviation change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 45 | 48 | 45
mg/dL | -20.1 (62.73) | -54.0 (67.51) | -40.9 (65.72)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0374, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided

14. Secondary Outcome: Mean Change in Post-prandial Insulin From Week 0(Baseline) to Week 16
Description: mean change in post-prandial insulin from Week 0(baseline) to week 16 with standard deviation change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 43 | 46 | 44
mg/dL | 3.898 (22.8717) | 1.962 (26.0326) | 4.832 (24.6608)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.2701, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.6117, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.2007, t-test, 2 sided

15. Secondary Outcome: Change in Low-Density Lipoprotein-C(LDL-C) From Week 0(Baseline) to Week 16 Least Squares Mean
Description: change in LDL-C from Week 0(baseline) to week 16 least squares mean with 95% confidence intervals change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 43 | 47 | 44
mg/dL | -19.5 [-26.5 to -12.6] | 4.9 [-1.8 to 11.5] | 6.2 [-0.7 to 13.0]

16. Secondary Outcome: Mean Change in LDL-C From Week 0(Baseline) to Week 16
Description: mean change in LDL-C from Week 0(baseline) to week 16 with standard deviation change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 43 | 47 | 44
mg/dL | -19.7 (23.85) | 5.5 (28.27) | 5.7 (22.33)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.1864, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0999, t-test, 2 sided

17. Secondary Outcome: Mean Percentage of Change in LDL-C Levels From Week 0(Baseline) to Week 16
Description: mean percent change in LDL-C levels from Week 0(baseline) to Week 16 mean with standard deviation change = week 16 - week 0.
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change in LDL-C
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 43 | 47 | 44
% change in LDL-C | -16.40 (19.443) | 7.41 (25.989) | 7.61 (21.180)
Statistical Analysis 1: Comparison: Colesevelam; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Rosiglitazone; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0566, t-test, 2 sided
Statistical Analysis 3: Comparison: Sitagliptin; P-value presents results from 1-sample t-test for within-treatment difference from baseline; Test type: Superiority or Other; p = 0.0217, t-test, 2 sided

18. Secondary Outcome: Mean Percentage of Change in LDL-C Levels From Week 0(Baseline) to Week 16 (Least Squares Mean)
Description: percent change in LDL-C levels from Week 0(baseline) to Week 16 (least squares mean with 95% confidence interval)
Time Frame: 16 weeks change = week 16 - week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: % change in LDL-C
Arm/Group | Colesevelam | Rosiglitazone | Sitagliptin
Number analyzed (Participants) | 43 | 47 | 44
% change in LDL-C | -16.24 [-22.68 to -9.81] | 6.92 [0.76 to 13.08] | 7.98 [1.62 to 14.34]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reflects the following restrictive language in the Clinical Study Agreements: "If identified by DSI, any of DSI's confidential information as defined herein shall be deleted…Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publication prepared by the Study Site."